CLINICAL TRIAL: NCT05244538
Title: Interest of Virtual Reality Distraction in the Management of Patients Benefiting From Oocyte Retrieval
Brief Title: Effectiveness of Hypnosis Via Virtual Reality During Oocyte Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYPNOFIV
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Virtual Reality Therapy; Fertilization in Vitro; Propofol; Remifentanil; Conscious Sedation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Distraction (Experimental): In the experimental group, patients will benefit from a 20-minute VR. Patients will watch a forest walk in virtual reality while listening to narrations designed to induce relaxation and meditation. If the oocyte retrieval was not completed within 20 minutes, patients will watch the same VR program again.The TCI remifentanil and propofol will be connected to the infusion but will be stopped and titrated if discomfort.
  Interventions: Device: Virtual reality distraction
- Sedation group (Active Comparator): Target controlled infusion (TCI) of remifentanil will be started at an effect concentration (Ce) of 1.5 ng/mL and TCI propofol at Ce 1.5 ug/mL.
  The concentration of remifentanil will be adjusted in 0.5 ng/ml increments based on hand sign from the patient with a maximum effect concentration of remifentanil at 2.5 ng/ml.
  The concentration of propofol will be adjusted by an effect concentration of 0.5 ug/ml with a maximum of 1.5 ug/ml, in this case according to a 5-point scale
  1. fully awake and oriented
  2. drowsy
  3. eyes closed, responds quickly to verbal commands
  4. eyes closed, aroused only by mild physical stimulation
  5. eyes closed, not aroused by mild physical stimulation) A sedation score of 3 will be the target throughout the procedure.
  Interventions: Drug: Propofol-remifentanil sedation

INTERVENTIONS:
Device: Virtual reality distraction — Patients will be exposed to a virtual reality representing a forest walk. A reduction of at least 50 percent in the remifentanil and propofol doses required for oocyte retrieval is expected.
  Arms: Virtual Reality Distraction
Drug: Propofol-remifentanil sedation — Target controlled infusion (TCI) of remifentanil will be started at an effect concentration (Ce) of 1.5 ng/mL and TCI propofol at Ce 1.5 ug/mL.
  The concentration of remifentanil will be adjusted in 0.5 ng/ml increments based on hand sign from the patient with a maximum effect concentration of remifentanil at 2.5 ng/ml.
  Arms: Sedation group

SUMMARY:
This study compares hypnosis via virtual reality to sedation with commonly used intravenous anesthetic agents (propofol and remifentanil) during oocyte retrieval.

The main objective of this prospective randomized controlled study will be a reduction of 50 percent of the doses of remifentanil and propofol administered during oocyte retrieval while maintaining satisfaction with the quality of care.

DETAILED DESCRIPTION:
Transvaginal ultrasound-guided oocyte retrieval is a fundamental step in the treatment of in vitro fertilization (IVF).

To date, no anesthetic technique has demonstrated superiority in terms of efficacy, tolerance or analgesia.

Virtual Reality Distraction has been studied for its clinical applications.

Patients will be included during the consultation with either the gynecologist or the anesthetist who will explain the protocol to the patient and give her consent to sign.

After obtaining their informed consent, the patient will be randomized into two groups based on a computer-generated randomization list (QuickCalcs program; GraphPad Software Inc) either into the experimental or in the control group.

In the experimental group, patients will benefit from a 20-minute virtual reality. Patients will watch a forest walk in virtual reality while listening to narrations designed to induce relaxation and meditation. If the oocyte retrieval was not completed within 20 minutes, the patient will watch the virtual reality program again. The target-controlled infusion of remifentanil and propofol will be connected to the patient, and only titrated to patient's comfort.

In the control group, patients will immediately benefit from an infusion of remifentanil and propofol titrated in a well-protocolized manner according to the patient's comfort.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients undergoing oocytes retrieval for in vitro fertilization

Exclusion Criteria:

* Presence of any psychiatric disorders
* Presence of a visual acuity disorder or hearing abnormality.
* Dementia
* Limited knowledge of French
* Diagnosis of balance disorders or epilepsy
* Claustrophobia
* Stage 4 endometriosis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patient undergoing in vitro fertilization
Enrollment: 48 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Dose reduction in propofol and remifentanil requirements | 2 hours
  Total dose of propofol (mg) and remifentanil (mcg) will be recorded in each group. A reduction of at least 50 percent of propofol and remifentanil doses will be expected in order to conclude on a superiority of the virtual reality distraction.

SECONDARY OUTCOMES:
Patient's comfort | 4 hours, during surgery
  Patient comfort will be measured using a five-point Gloucester Comfort scale ranging from 1 (comfortable) to 5 (severe discomfort)

CONTACTS AND LOCATIONS:
Overall Officials: Turgay Tuna, MD, PhD, Study Director — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Belgium